CLINICAL TRIAL: NCT02866214
Title: Evaluation of the Effect of Febuxostat on Endothelial Dysfunction in Hemodialysis Patients.
Brief Title: Effect of Febuxostat on Endothelial Dysfunction in Hemodialysis Patients.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona AlShahawey AlSayed Ghazy, Administrator at clinical pharmacy department ., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: phCL 35
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Endothelial Dysfunction; Endstage Renal Disease
MeSH Terms: interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Group I (Experimental): This Group of Patients will receive Febuxostat Drug along with their Standard Treatment.
  Interventions: Drug: Febuxostat
- Group II (Placebo Comparator): This Group of Patients will receive Placebo along with their standard Treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat — Film Coated Tablets of Donifoxate (Eva Pharma company ) 40mg administered thrice weekly post hemodialysis session
  Other Names: Donifoxate
  Arms: Group I
Drug: Placebo — Film Coated Tablets (Placebo) to be administered thrice weekly post hemodialysis session.
  same color, taste , size . Same all ingredients except Febuxostat (Active ingredient) .
  Arms: Group II

SUMMARY:
The Purpose of this study is to determine if the Febuxostat has an effect on endothelial dysfunction on hemodialysis patients.

DETAILED DESCRIPTION:
Aim of The Work:

1- Evaluation of the effect of febuxostat on endothelial dysfunction in hemodialysis patients, through detection of:

1. Primary endpoint:

   • Reduction in Asymmetrical Dimethylarginine (ADMA)
2. Secondary endpoints:

   * Assessing the change in serum High sensitivity C-reactive protein (hsCRP)
   * Assessing the change in serum Uric acid - The criteria for inclusion:

     1. Outpatients on maintenance hemodialysis.
     2. Age from 18-70 years old.
     3. Serum UA level 7.0 mg/dL or more.
     4. Stable clinical condition (no hospitalization in the previous 3 months)

The exclusion criteria:

1. Current urate-lowering therapy. (allopurinol, probenecid, bucolome, febuxostat)
2. History of hypersensitivity to febuxostat.
3. Current treatment with mercaptopurine, azathioprine, pyrazinamide, or ethambutol.
4. Participant in an another clinical trial within the past 4 weeks.
5. Judged to be unsuitable as a subject by the attending physician.

After two months , the patient will be reassessed regarding:

A. ADMA serum level. B. Change in serum hsCRP. C. Change in serum Uric acid level.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients on maintenance hemodialysis.
* Age from 18-70 years old.
* Serum Uric Acid level 7.0 mg/dL or more.
* Stable clinical condition (no hospitalization in the previous 3 months)
* Informed consent in accordance with the Declaration of Helsinki.

Exclusion Criteria:

* Current urate-lowering therapy. (allopurinol, probenecid, bucolome, febuxostat)
* History of hypersensitivity to febuxostat.
* Current treatment with mercaptopurine, azathioprine, pyrazinamide, or ethambutol.
* Participant in an another clinical trial within the past 4 weeks.
* Judged to be unsuitable as a subject by the attending physician

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Asymmetric Dimethylarginine physiological marker | 2 months
  Asymmetric dimethylarginine (ADMA) physiological marker for assessing endothelial dysfunction will be measured for all the anticipated 50 patients at time zero and by the end of the two months.

SECONDARY OUTCOMES:
Uric Acid , physiological parameter | 2 months
  Uric acid,physiological parameter for assessing the grade of hyperuricemia will be measured for all the anticipated 50 patients at time zero and by the end of the two months.
High sensitivity C-reactive protein physiological marker | 2 months
  HsCRP , physiological marker for assessing inflammation will be measured for all the anticipated 50 patients at time zero and by the end of the two months.